CLINICAL TRIAL: NCT02945202
Title: Einfluss Der Trabekulektomie Und Der Kombinierten Phako-Trabekulektomie Auf Den Kornealen Astigmatismus
Brief Title: Influence of Trabeculectomy and Phaco-trabeculectomy on Corneal Astigmatism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Astigmatismus2017
Record Dates: First submitted 2016-10-20; First posted 2016-10-26 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Astigmatism; Glaucoma
MeSH Terms: conditions — Astigmatism; Glaucoma | interventions — Biometry; Refraction, Ocular; Corneal Topography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All Eyes (Other): All eyes undergo the same interventions. These are the following examinations: Biometry, Refraction and Corneal Topography. The examinations take place 6 months after surgery
  Interventions: Device: Biometry; Device: Refraction; Device: Corneal Topography

INTERVENTIONS:
Device: Biometry — All patients undergo all three examinations (biometry, refraction and corneal topography) 6 months after surgery
Device: Refraction — All patients undergo all three examinations (biometry, refraction and corneal topography) 6 months after surgery
Device: Corneal Topography — All patients undergo all three examinations (biometry, refraction and corneal topography) 6 months after surgery

SUMMARY:
This study investigates the effects of trabeculectomy and combined phacoemulsification plus trabeculectomy on corneal astigmatism.

DETAILED DESCRIPTION:
Prospectively, consecutive patients at the University Hospital of Zurich undergoing either trabeculectomy (trab) or phaco-trabeculectomy (phaco-trab) are included in this study between January and December 2017. The study interventions takes place 6 months after surgery and include examination of refraction, biometry and corneal topography in order to assess the patient's astigmatism. The values are compared to the preoperative baseline values, which are available from patient records.

ELIGIBILITY:
Inclusion Criteria:

* Trabeculectomy or Phaco-Trabeculectomy between 01/2017 and 12/2017
* Age ≥18 years

Exclusion Criteria:

* Acute or chronic corneal diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Difference in Astigmatism [Diopters (dpt)] | preoperative astigmatism compared to 6 months postoperatively

IPD SHARING:
Plan to Share IPD: No